CLINICAL TRIAL: NCT03119610
Title: The Physiologic Effects of Intranasal Oxytocin on Sarcopenic Obesity
Acronym: INOSO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sara Espinoza (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); The University of Texas Health Science Center, Houston (Other); The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor-Investigator, Sara Espinoza, Associate Professor of Medicine, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HSC20160661H
Record Dates: First submitted 2017-03-22; First posted 2017-04-18 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Sarcopenic Obesity; Sarcopenia; Aging; Sedentary Lifestyle
MeSH Terms: conditions — Obesity; Sarcopenia; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin nasal spray (Experimental): Oxytocin (Syntocinon), intranasal, 24IU, 4x a day for 8 weeks, self administered
  Interventions: Drug: Oxytocin nasal spray
- Placebo nasal spray (Experimental): Placebo nasal spray, 4x a day for 8 weeks, self administered
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Self administered Oxytocin nasal spray q.i.d. for 8 weeks versus placebo (normal saline nasal spray)
  Other Names: Intranasal oxytocin; Syntocinon nasal spray
  Arms: Oxytocin nasal spray
Drug: Placebo nasal spray — Self administered Placebo nasal spray q.i.d. for 8 weeks (normal saline nasal spray)
  Other Names: Saline nasal spray
  Arms: Placebo nasal spray

SUMMARY:
Obesity is highly prevalent in older adults and is a major cause of sarcopenia and disability in older adults. Although exercise can counteract the effects of obesity and sarcopenia, many have difficulty adhering to an exercise program and the benefits of exercise are variable. Therefore, there is an urgent need to test novel pharmacologic interventions to prevent disability and loss of independence. Oxytocin is a pituitary hormone released during parturition and lactation that is also known to suppress appetite in rodents and humans; and, recent small studies have found that intranasal oxytocin reduces body weight in adults. We propose a pilot study of intranasal oxytocin as a novel approach to promote weight loss and increase muscle mass in older subjects with sarcopenic obesity.

DETAILED DESCRIPTION:
The pilot study will be conducted at 3 sites in 9 visits over a period of 12+ weeks. Older sedentary subjects will be screened for sarcopenic obesity using a modified consensus definition and evaluated at baseline for safety labs, glucose tolerance, body composition, cognition and physical performance, as well as systemic inflammatory markers in blood and muscle tissue.

Eligible subjects self-administer 24 IU intranasal oxytocin four times a day for 8 weeks.

The study will examine whether the intervention will promote weight loss and preserve muscle mass, thereby preserving and/or improving physical function in older subjects with sarcopenic obesity.

Generalized linear mixed effects model will be used to evaluate the effect of oxytocin on the change of each continuous measure. The effect of oxytocin will be assessed by whether the time by oxytocin interaction is significantly different from 0 with a 2-sided p-value<0.05.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40 kg/m2
* Sedentary (< 2 strenuous exercise/week)
* Gait speed < 1 meter/second

Exclusion Criteria:

* Diabetes (ADA criteria)
* Heart disease (MI or New York Heart Classification grade III-IV)
* Poorly controlled hypertension (SBP > 170 or DBP >95 mm/Hg)
* Anemia (Hematocrit <34%)
* Renal Disease (Serum Creatinine >1.4, abnormal serum sodium levels, abnormal urinalysis, or physical exam findings indicative of fluid imbalance; individuals with underlying disorder of sodium/water balance, such as SIADH, diabetes insipidus, or psychogenic polydipsia)
* Liver Disease (AST/ALT/AlkPhos > 2x upper limit of normal)
* Use of systemic steroid, androgens, or anti-coagulants
* Active/unstable conditions: inflammatory, thyroid, autoimmune, gastrointestinal (GI), hematologic, or neoplastic disorders
* Individuals with underlying seizure disorder or underlying neurologic disorder that increases seizure risk
* Cognitive impairment (MiniCog <3), unstable mental illness, substance abuse, or history of eating disorder

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Espinoza, MD, Principal Investigator — The University of Texas Health Science Center, San Antonio
Locations (1):
- Texas Diabetic Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Espinoza SE, Lee JL, Wang CP, Ganapathy V, MacCarthy D, Pascucci C, Musi N, Volpi E. Intranasal Oxytocin Improves Lean Muscle Mass and Lowers LDL Cholesterol in Older Adults with Sarcopenic Obesity: A Pilot Randomized Controlled Trial. J Am Med Dir Assoc. 2021 Sep;22(9):1877-1882.e2. doi: 10.1016/j.jamda.2021.04.015. Epub 2021 May 21. PMID 34029521

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Started | 13 | 10
Completed | 12 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Customized [Count of Participants; unit: Participants] — Participants are included if age 60 or over.
  Participants
    Age, 60 or over | 13 | 10 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Intranasal oxytocin will promote weight loss and preserve muscle mass
Time Frame: Baseline to 8 weeks
Population: Two participants withdrew after randomization; 1 in Oxytocin and 1 in Placebo group. Data from these two subjects were not collected.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
Kilograms | 0.54 (1.6) | 0.04 (2.5)

2. Secondary Outcome: Change in Fat Mass
Description: Pre- and post-measurements of fat mass by dual energy x-ray absorptiometry (DXA) will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
Kilograms | -0.2 (0.99) | -0.1 (0.92)

3. Secondary Outcome: Change in Body Mass Index
Description: Pre- and post-measurements of lean mass by DXA will be examined for individual change with intranasal oxytocin. Change in body mass index (BMI).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
kg/m2 | 36.8 (3.5) | 36.8 (3.6)

4. Secondary Outcome: Change in Glucose Levels Measured Using the Glucose Tolerance Test
Description: Pre- and post-measurements of oral glucose tolerance test for 2-hour plasma glucose will be examined for individual change with intranasal oxytocin
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
mg/dL
  Fasting glucose | 3.36 (10.18) | 2.85 (6.28)
  2-hour glucose | -3.15 (31.126) | -3.375 (14.88)

5. Secondary Outcome: Change in Short Physical Performance Battery (SPPB)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin. This battery of tests is scored on a scale with 3 SPPB calculation components:
  1. Ability to stand for 10 seconds with feet in 3 different positions, scored from 0 min to 4 maximum, with a higher score indicating better balance.(3 Balance subsets: side by side stand scored from 0-1; semi-tandem stance scored from 0-1; tandem stance scored from 0-2)
  2. Two timed trials of a 3m or 4 m walk (fastest recorded). Scoring is from 0-4, with 0 being unable to walk and 4 indicating a faster walk time.
  3. Time to rise from a chair five times is scored from 0-4, with 0 being unable to complete the activity, and 4 indicating that time to complete is less than 11.1 seconds.
  Total Score is the sum of all 3 scores: Minimum = 0 Maximum = 12. Higher scores indicate better lower extremity function.
  Difference between baseline and 8 week performance is reported.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
score on a scale | 0.5 (1.446) | 0.625 (1.598)

6. Secondary Outcome: Change in HbA1c (Hemoglobin A1c)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
Percentage | -0.05 (0.1857) | 0.286 (0.1254)

7. Secondary Outcome: Change in Waist Circumference
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: centimeteres
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
centimeteres | -0.6958 (4.8662) | -1.373 (2.1997)

8. Secondary Outcome: Change in Total Cholesterol
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
mg/dL | -11.18 (17.417) | -1.143 (16.056)

9. Secondary Outcome: Change in Low Density Lipoproteins (LDL)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
mg/dL | -8.727 (16.224) | 4.1429 (11.539)

10. Secondary Outcome: Change in High Density Lipoproteins (HDL)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
mg/dL | 1.000 (2.8983) | 0.1429 (3.8408)

11. Secondary Outcome: Change in Triglycerides
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
mg/dL | -16.82 (23.828) | -26.29 (46.903)

12. Secondary Outcome: Change in Center for Epidemiologic Studies Scale (CES-D)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin. This is measured on a 20 item scale using the following scoring using number of week days:
  1. Rarely or none of the time ( less than 1 day)
  2. Some or a little of the time (1-2 days)
  3. Occasionally or a moderate amount of time (3-4 days)
  4. Most or all of the time (5-7 days) SCORING: zero for answers =1), 1 for answers =2), 2 for answers =3) column, 3 for answers =4) The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
score on a scale | -1.375 (2.1860) | 0.2222 (2.7285)

13. Secondary Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: Pre- and post-measurements will be examined for individual change with intranasal oxytocin. A 30-point test, with a score of 0 or 1 assigned to each item. The minimum score is 0 and the maximum is 30. The higher the score, the less cognitive impairment.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 12 | 9
score on a scale | 1.0000 (1.5954) | 0.4444 (1.3333)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 12/12 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin Nasal Spray (N=12) | Placebo Nasal Spray (N=9)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tiredness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Lightheaded (Nervous system disorders) | 2 (2) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Bruise related to biopsy (Vascular disorders) | 1 (1) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms, hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms, legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Throat itching (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Loose stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased bowel movement (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bladder disturbance (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03119610/Prot_SAP_000.pdf